CLINICAL TRIAL: NCT06202820
Title: CV CARE: CardioVascular Care of Androgen Related Effects in Prostate Cancer Patients
Brief Title: CV CARE: CardioVascular Care in PC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Alicia Morgans, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-311
Record Dates: First submitted 2024-01-01; First posted 2024-01-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Cardiovascular Diseases
Keywords: Prostate Cancer; Cardiovascular Diseases; Cardiovascular Risk
MeSH Terms: conditions — Prostatic Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CV Care Program (Experimental): Study procedures will be conducted as follows:
  * Standard of care androgen deprivation therapy.
  * 4 week standard-of-care follow up visit in clinic with CV care education module completion.
  * 12-week standard-of-care prostate cancer care visit with oncologist.
  * 24-week standard-of-care post-ADT visit in clinic with CV Care module completion, surveys, and exit interview with clinical team members.
  * The CV Care program will be revised through participant feedback from assessments, surveys, focus groups, and exit-interviews. The revised CV Care Program will be used in the next cohort.
  Interventions: Behavioral: CV Care Program
- CV Care Program 2 (Experimental): Study procedures will be conducted as follows:
  * Standard of care androgen deprivation therapy.
  * 4 week standard-of-care follow up visit in clinic with CV care education module completion.
  * 12-week standard-of-care prostate cancer care visit with oncologist.
  * 24-week standard-of-care post-ADT visit in clinic with CV Care module completion, surveys, and exit interview with clinical team members.
  * Participant feedback from surveys, exit-interviews, and possibly focus groups will be collected.
  Interventions: Behavioral: CV Care Program

INTERVENTIONS:
Behavioral: CV Care Program — Comprised of two, in-clinic, counseling sessions with oncology nurse practitioner or physician assistant for education on cardiovascular disease (CVD) and cardiovascular risk factors as well as recommendations for management.

SUMMARY:
This research is being done to test a program to assess and manage reversible cardiovascular (CV) risk factors in participants with prostate cancer starting androgen deprivation therapy (ADT), with the goal of integrating a standardized method into Dana-Farber Cancer Institute clinics for all such participants.

The name of the intervention used in this research study is:

CV Care (cardiovascular risk assessment and management program)

DETAILED DESCRIPTION:
This research is being done to test a program to assess and manage reversible cardiovascular (CV) risk factors in participants with prostate cancer starting androgen deprivation therapy (ADT), with the goal of integrating a standardized method into Dana-Farber Cancer Institute clinics for all such participants.

Study procedures including screening for eligibility, treatment visits, questionnaires and surveys, and blood and urine tests.

Participation in this research study is expected to last about 6 months.

It is expected that about 60-150 people will take part in this study.

This study is supported by the National Comprehensive Cancer Network (NCCN) through grant funding provided by Pfizer Myovant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologic diagnosis of prostate adenocarcinoma. Participants with any stage of prostate cancer are eligible, as long as treatment with at least 24 weeks of ADT is recommended by their treating physician.
* Participants must have been prescribed a plan for treatment with at least 24 weeks of ADT, and can have received up to 12 weeks of ADT therapy.
* Participants must be willing to participate in two CV CARE visits at weeks 12 and 24 after ADT initiation.
* Participants must be willing to have their follow up visits for ADT management at DFCI Longwood site.
* Participants must be willing to undergo lab and blood pressure assessments, which can include local labs and home blood pressure checks if they wish to do virtual visits for follow up care.
* Participants can have pre-existing CVD and/or CV risk factors, but this is not a requirement for inclusion.
* Participants receiving combination treatment with an androgen receptor signaling inhibitory, some examples being (abiraterone acetate, enzalutamide, darolutamide, apalutamide, or bicalutamide), immunotherapy (pembrolizumab), or PARP inhibitor (olaparib, rucaparib) are eligible.
* Age ≥18 years.
* Life expectancy of greater than 6 months.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of major adverse cardiac event, including myocardial infarction, new congestive heart failure (CHF) or CHF exacerbation, or stroke, within the past 24 weeks due to complicated comorbidities that necessitate close collaboration between the participant and their cardiologist.
* Participants who have already been on ADT therapy for more than 12 weeks are ineligible due to their treatment cycle being incompatible with the quality improvement initiative's trial design. ADT therapy is defined as either a GnRH agonist or antagonist.
* Participants receiving combination treatment with ADT and chemotherapy (docetaxel, cabazitaxel, carboplatin), radioligand therapy (radium-223, 177PSMA-lutetium-617), or treatment on a clinical trial are not eligible due to potential for more intensive symptom management that may be required for optimal support of their cancer-directed treatment.
* Participants actively included in therapeutic clinical trials are not eligible due to their greater time constraints.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant Retention Rate in CV CARE 2 | Weeks 4 and 24 in CV CARE 2
  The percentage of a continued participation rate at week 24 of participants who participate at week 4 in the revised iteration of the program (CV CARE 2).

SECONDARY OUTCOMES:
Proportion of Participants on Statin Medications in CV CARE | 5 months (From 4 weeks after ADT initiation to the week 24 on-treatment visit)
  The percentage of participants who initiate or adjust statin medication usage during the period between 4 weeks after ADT initiation and the week 24 on-treatment visit among individuals with ASCVD risk scores exceeding 10% and 20% at week 4 of the study.
Proportion of Participants on Statin Medications in CV CARE 2 | 5 months (From 4 weeks after ADT initiation to the week 24 on-treatment visit)
  The percentage of participants who initiate or adjust statin medication usage during the period between 4 weeks after ADT initiation and the week 24 on-treatment visit among individuals with ASCVD risk scores exceeding 10% and 20% at week 4 of the study.
Proportion of Participants on Blood Pressure Medications in CV CARE | 5 months (From 4 weeks after ADT initiation to the week 24 on-treatment visit)
  The percentage of participants who initiate or adjust blood pressure medication usage during the period between 4 weeks after ADT initiation and the week 24 on-treatment visit among individuals with ASCVD risk scores exceeding 10% and 20% at week 4 of the study.
Proportion of Participants on Blood Pressure Medications in CV CARE 2 | 5 months (From 4 weeks after ADT initiation to the week 24 on-treatment visit)
  The percentage of participants who initiate or adjust blood pressure medication usage during the period between 4 weeks after ADT initiation and the week 24 on-treatment visit among individuals with ASCVD risk scores exceeding 10% and 20% at week 4 of the study.
Proportion of Participants with Blood Pressure Below 130/85 (mmHg) in CV CARE | 6 months (From the ADT initiation to the week 24 on-treatment visit)
  The comparison of proportion of participants with a blood pressure below 130/85 mmHg between the average blood pressure levels of weeks 12 and 24 of the program and the average blood pressure levels of ADT initiation and week 4.
Proportion of Participants with Blood Pressure Below 130/85 (mmHg) in CV CARE 2 | 6 months (From the ADT initiation to the week 24 on-treatment visit)
  The comparison of proportion of participants with a blood pressure below 130/85 mmHg between the average blood pressure levels of weeks 12 and 24 of the program and the average blood pressure levels of ADT initiation and week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Morgans, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu